CLINICAL TRIAL: NCT03267966
Title: Margin Status After Pancreaticoduodenectomy for Cancer. Results of a Multicentric Prospective Randomized Trial
Brief Title: Margin Status After Pancreaticoduodenectomy for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Collaborators: Humanitas Hospital, Italy (Other); Azienda Ospedaliero, Universitaria Pisana (Other); Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Gennaro Nappo, M.D., Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NI 01/13
Record Dates: First submitted 2017-08-11; First posted 2017-08-31 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cancer; Cholangiocarcinoma; Ampullary Cancer
Keywords: periampullary cancer; margin status; R1 resection; clearance margin
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Leeds Pathology Protocol (LEEPP)
  Interventions: Diagnostic Test: Leeds Pathology Protocol (LEEPP)
- Group B (No Intervention): "Conventional" method of pathological evaluation

INTERVENTIONS:
Diagnostic Test: Leeds Pathology Protocol (LEEPP) — LEEPP includes: 1) multicolor inking; 2) axial slicing; 3) circumferential margin; 4) 1-mm clearance
  Arms: Group A

SUMMARY:
This multicentric prospective randomized controlled trial (RCT) compares the Leeds Pathology Protocol (LEEPP) with other "conventional" pathological protocol of PD specimen for periampullary cancer. Our aims were to evaluate the impact of the protocol and of the clearance on R1 rate and its prognostic value.

ELIGIBILITY:
Inclusion Criteria:

* pancreaticoduodenectomy for periampullary cancer

Exclusion Criteria:

* diagnosis of neuroendocrine neoplasm;
* previous pancreatic surgery;
* frozen section of each transection margins not performed or presence of positive transection margins without further resection (R1 intraoperative resection);
* presence of macroscopic residual tumor (R2 resection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
R1 resection rate | 1 month
  To evaluate difference in terms of R1 resection rates between study groups with 0-mm and 1-mm clearance

SECONDARY OUTCOMES:
pathological data | 1 month
  To evaluate differences in pathological results (T status, N status, number of blocks, number of lymphnodes, etc) between the two study groups
oncological results | 60 months
  To evaluate the correlation between R1 resection and oncological results (local recurrence, overall survival) in the two study groups

IPD SHARING:
Plan to Share IPD: No